CLINICAL TRIAL: NCT05759403
Title: Comparative Study Between Parkinson's Disease and Parkinson Dementia Complex : Genetics, Clinical, Neurophysiological
Brief Title: Comparison Between Parkinson's Disease and Parkinson's Dementia Complex (Genetically,Clinical and Electrophysiological)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor doctor, Assiut University
Other Study IDs: TMS in Parkinson's
Record Dates: First submitted 2023-02-02; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease Dementia; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for genetic analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with parkinson's disease: Genetic analysis, clinical data , cortical excitbility
  Interventions: Diagnostic Test: Cortical excitability using transcranial magnetic stimulation
- patients with Parkinson dementia complex: Genetic analysis, clinical data , cortical excitbility
  Interventions: Diagnostic Test: Cortical excitability using transcranial magnetic stimulation

INTERVENTIONS:
Diagnostic Test: Cortical excitability using transcranial magnetic stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive neurophysiological technique for assessing human motor cortical function. With TMS, the underlying motor cortex is stimulated by an electric current induced by a transient magnetic field, generated in response to the passage of a large current through the stimulating coil located on the patient's scalp.

SUMMARY:
To compare between Idiopathic PD versus Parkinson-Dementia complex using different modalities: Demographic, Clinical, genetic, Psychometric and electrophysiologically

DETAILED DESCRIPTION:
Parkinson's disease (PD), is one of the commonest neurodegenerative disorders with a severe progressive course and major impact on patients' quality of life. The development of late-onset PD likely results from the interaction of genetic and environmental factors in the context of brain aging.

Although several environmental exposures have been implicated, evidence for their causal contributions is limited.

PD in Egypt is a rapidly emerging concern as prevalence rose by 40.7% between 1990 and 2016, one of the highest increases in the world. which influences us to dig further in the genetic basis behind the scenes leading to that leap.

Cognitive impairment in PD constitutes a major source of disease burden for patients and families, and has a significant negative effect on patients' quality of life. Cognitive impairment without dementia is designated as mild cognitive impairment of PD (PD-MCI), where the activities of daily living are grossly preserved, whereas dementia associated with PD is designated as PD-D.

Parkinson's disease dementia is a neurofibrillary tangle degeneration involving the deposition of Alzheimer-type tau, predominantly in the mesial temporal cortex, brainstem, and basal ganglia.

The prevalence of Parkinson's Disease Dementia (PD-D) in the general population aged 65 years and over was 0.3 to 0.5%, and 3 to 4% of patients with dementia in the general population were estimated to be due to PD-D.

Transcranial magnetic stimulation (TMS) is a noninvasive neurophysiological technique for assessing human motor cortical function. With TMS, the underlying motor cortex is stimulated by an electric current induced by a transient magnetic field, generated in response to the passage of a large current through the stimulating coil located on the patient's scalp.

ELIGIBILITY:
Inclusion Criteria:

* All participants must fulfill the following inclusion criteria of UINTED KINGDOM bank criteria of PD Men or women of at least 50-80 years of age.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow up.
* Medically stable outpatients with confirmed diagnosis of idiopathic PD according to United Kingdom Brain Bank Criteria
* Clear written informed consent from each participant in the trial.
* Patients after at least 6 h free of parkinsonian drugs (off-state).
* For the Parkinson's Dementia Complex group, dementia must be evident through history taking or clinical examination

Exclusion Criteria:

* Pregnants, breastfeeding, or willing to be pregnant during the study.
* Presence of clinically significant medical or psychiatric condition that may increase the risk associated with the study
* Participation in any other type of medical research that may interfere with the interpretation of the study.
* Patients with severe motor disability (bed-ridden ) that may interfere with the study procedure.
* History of surgical or invasive intervention for Parkinson disease.
* Patients with history of seizures or epilepsy including history in a first degree relative or patients on treatment that reduce seizure threshold.
* For the Parkinson's Dementia Complex group, Subject with dementia due to other diseases or with Parkinson's dementia complex and contribution of other disorders (Mixed dementia)
* Brain imaging suggesting another diagnosis.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with parkinson's disease and parkinson dementia complex
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Score on MDS-UPDRS | through study completion, an average of 1 year
  Score on MDS-UPDRS
Score on mini mental state examination | through study completion, an average of 1 year
  Score on mini mental state examination

SECONDARY OUTCOMES:
Score on PDQ-39 | through study completion, an average of 1 year
  Score on PDQ-39
Score on Score on Montreal Cognitive Assessment | through study completion, an average of 1 year
  Score on Score on Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen H, Ritz B. The Search for Environmental Causes of Parkinson's Disease: Moving Forward. J Parkinsons Dis. 2018;8(s1):S9-S17. doi: 10.3233/JPD-181493. PMID 30584168
- [Background] Ball N, Teo WP, Chandra S, Chapman J. Parkinson's Disease and the Environment. Front Neurol. 2019 Mar 19;10:218. doi: 10.3389/fneur.2019.00218. eCollection 2019. PMID 30941085
- [Background] Priyadarshi A, Khuder SA, Schaub EA, Priyadarshi SS. Environmental risk factors and Parkinson's disease: a metaanalysis. Environ Res. 2001 Jun;86(2):122-7. doi: 10.1006/enrs.2001.4264. PMID 11437458
- [Background] Bellou V, Belbasis L, Tzoulaki I, Evangelou E, Ioannidis JP. Environmental risk factors and Parkinson's disease: An umbrella review of meta-analyses. Parkinsonism Relat Disord. 2016 Feb;23:1-9. doi: 10.1016/j.parkreldis.2015.12.008. Epub 2015 Dec 17. PMID 26739246
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Sezgin M, Bilgic B, Tinaz S, Emre M. Parkinson's Disease Dementia and Lewy Body Disease. Semin Neurol. 2019 Apr;39(2):274-282. doi: 10.1055/s-0039-1678579. Epub 2019 Mar 29. PMID 30925619
- [Background] Morris HR, Steele JC, Crook R, Wavrant-De Vrieze F, Onstead-Cardinale L, Gwinn-Hardy K, Wood NW, Farrer M, Lees AJ, McGeer PL, Siddique T, Hardy J, Perez-Tur J. Genome-wide analysis of the parkinsonism-dementia complex of Guam. Arch Neurol. 2004 Dec;61(12):1889-97. doi: 10.1001/archneur.61.12.1889. PMID 15596609
- [Background] Aarsland D, Zaccai J, Brayne C. A systematic review of prevalence studies of dementia in Parkinson's disease. Mov Disord. 2005 Oct;20(10):1255-63. doi: 10.1002/mds.20527. PMID 16041803
- [Background] Chen R, Cros D, Curra A, Di Lazzaro V, Lefaucheur JP, Magistris MR, Mills K, Rosler KM, Triggs WJ, Ugawa Y, Ziemann U. The clinical diagnostic utility of transcranial magnetic stimulation: report of an IFCN committee. Clin Neurophysiol. 2008 Mar;119(3):504-532. doi: 10.1016/j.clinph.2007.10.014. Epub 2007 Dec 11. PMID 18063409
- [Background] Rossini PM, Barker AT, Berardelli A, Caramia MD, Caruso G, Cracco RQ, Dimitrijevic MR, Hallett M, Katayama Y, Lucking CH, et al. Non-invasive electrical and magnetic stimulation of the brain, spinal cord and roots: basic principles and procedures for routine clinical application. Report of an IFCN committee. Electroencephalogr Clin Neurophysiol. 1994 Aug;91(2):79-92. doi: 10.1016/0013-4694(94)90029-9. No abstract available. PMID 7519144
- [Background] Ziemann U, Netz J, Szelenyi A, Homberg V. Spinal and supraspinal mechanisms contribute to the silent period in the contracting soleus muscle after transcranial magnetic stimulation of human motor cortex. Neurosci Lett. 1993 Jun 25;156(1-2):167-71. doi: 10.1016/0304-3940(93)90464-v. PMID 8414181
- [Background] Chen R, Lozano AM, Ashby P. Mechanism of the silent period following transcranial magnetic stimulation. Evidence from epidural recordings. Exp Brain Res. 1999 Oct;128(4):539-42. doi: 10.1007/s002210050878. PMID 10541749
- [Background] Daskalakis ZJ, Christensen BK, Chen R, Fitzgerald PB, Zipursky RB, Kapur S. Evidence for impaired cortical inhibition in schizophrenia using transcranial magnetic stimulation. Arch Gen Psychiatry. 2002 Apr;59(4):347-54. doi: 10.1001/archpsyc.59.4.347. PMID 11926935